CLINICAL TRIAL: NCT00462280
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Trial of Lovastatin for Various Endpoints of Melanoma Pathobiology
Brief Title: Lovastatin in Treating Patients At High Risk of Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NCI-2009-00896; NCI-2009-00896 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2006-4937; UCI03-1-01; CDR0000540141; UCI 06-06 (Other: Chao Family Comprehensive Cancer Center); UCI03-1-01 (Other: DCP); N01CN35160 (NIH)
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Results first posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-02

CONDITIONS: Precancerous Condition; Stage 0 Melanoma; Stage I Melanoma; Stage II Melanoma
MeSH Terms: conditions — Precancerous Conditions; Melanoma | interventions — Lovastatin; Biopsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Two matched nevi group - Lovastatin (Experimental): Patients with two matched nevi received lovastatin PO QD for up to 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lovastatin; Procedure: biopsy; Procedure: laboratory biomarker analysis
- Two Matched Nevi Group - Placebo (Placebo Comparator): Patients with two matched nevi received placebo PO QD for up to 6 months in the absence of disease progression or unacceptable toxicity
  Interventions: Other: placebo; Procedure: biopsy; Procedure: laboratory biomarker analysis
- One large nevi group - Lovastatin (Experimental): Patients who have one large nevi received lovastatin PO QD for up to 6 months in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: lovastatin; Procedure: biopsy; Procedure: laboratory biomarker analysis
- One Large Nevi Group - Placebo (Placebo Comparator): Patients who have one large nevi received placebo PO QD for up to 6 months in the absence of disease progression or unacceptable toxicity
  Interventions: Other: placebo; Procedure: biopsy; Procedure: laboratory biomarker analysis

INTERVENTIONS:
Drug: lovastatin — Given PO
  Other Names: Lovastatin Sodium; Mevacor; Mevinolin; Monacolin K
  Arms: One large nevi group - Lovastatin; Two matched nevi group - Lovastatin
Other: placebo — Given PO
  Other Names: PLCB
  Arms: One Large Nevi Group - Placebo; Two Matched Nevi Group - Placebo
Procedure: biopsy — Correlative studies
  Other Names: biopsies
Procedure: laboratory biomarker analysis — Correlative studies

SUMMARY:
The use of lovastatin may slow disease progression in patients at high risk of melanoma. It is not yet known whether lovastatin is more effective than a placebo in treating patients at high risk of melanoma. This randomized phase II trial studies how well giving lovastatin or placebo works in treating patients at high risk of melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the primary endpoint of the trial, by analysis of histopathologic regression of atypical nevi in response to a 6-month trial of oral (PO) lovastatin vs. placebo in subjects with atypical nevi.

SECONDARY OBJECTIVES:

I. To evaluate clinical regression of atypical nevi in the lovastatin vs. placebo group.

II. To evaluate the secondary endpoint of changes in nevi numbers on subjects' backs in the lovastatin vs. placebo groups.

III. To evaluate a number of molecular biomarkers as secondary endpoints in the lovastatin vs. placebo groups.

IV. To evaluate the correlation of serum markers known to be affected by lovastatin with the endpoints chosen above.

V. To evaluate the safety and tolerability of the dosing regimen, and the dose escalation.

OUTLINE: Patients are randomized into 1 of 2 treatment arms per group.

ARM I: Patients (with two matched nevi OR one large nevi) receive lovastatin PO once daily (QD) for up to 6 months in the absence of disease progression or unacceptable toxicity.

ARM II: Patients (with two matched nevi OR one large nevi) receive placebo PO QD for up to 6 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least 2 clinically atypical nevi on the body that are reasonably matched in regards to level of clinical atypia, or one atypical mole and another atypical mole >= 8 mm in diameter (for this pair the two moles do not have to be closely matched and only one of them must be >= 8 mm in diameter)
* A history of melanoma is not required for study entry
* Patients with completely resected stage I or II who have not received adjuvant therapy in the past 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 1 or better (Karnofsky > 70%)
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 X within normal limits
* Creatinine within normal institutional limits
* Ability to understand and the willingness to sign the written informed consent
* Subjects willing and able to participate for the full duration of the study
* For women of child-bearing potential (women are considered not of childbearing potential if they are at least 2 years post-menopausal and/or surgically sterile), she:

  * has been using adequate contraception (abstinence, intrauterine device [IUD], birth control pills, or spermicidal gel with diaphragm or condom) since her last menses and will use adequate contraception during the study
  * is not lactating, and
  * has had a documented negative serum pregnancy test within 30 days prior to the first dose of study medication Should a woman become pregnant or suspect she is pregnant while participating in this study, she will be taken off study and be advised to inform her treating physician immediately; a telephone follow-up with the subject post-delivery will be completed to obtain outcome of pregnancy
* Men partnered with a female of child-bearing age must agree to use adequate contraception while on the study (i.e. abstinence, IUD, birth control pills, or spermicidal gel with diaphragm or condom)

Exclusion Criteria:

* Subjects with untreated melanoma of any stage or locally advanced (>= 4 mm in Breslow's thickness) or metastatic (stage III or IV) melanoma; subjects with melanoma may be considered for trial after complete resection of Stage I or II melanoma and those who have declined or are ineligible to go on any available adjuvant clinical trials known to the investigators or the subjects are eligible
* Subjects who are on adjuvant therapy or experimental therapy for melanoma currently or within the last 3 months prior to enrollment into this study
* Subjects currently or within the last three months before enrollment on lipid lowering agents of any type
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lovastatin
* Clinically significant unrelated systemic illness
* Subjects with any medical or psychosocial condition that, in the opinion of the investigator, could jeopardize his/her participation in and compliance with the study
* Subjects may not be receiving any other investigational agents
* Pregnant or breast feeding females, or females of child bearing age not using a reliable method of contraception (use of lovastatin is contraindicated in pregnancy)
* Subjects who have been diagnosed with malignancies other than cutaneous melanoma, cutaneous basal cell carcinoma, or cutaneous squamous cell carcinoma within 5 years of study entry, unless they:

  * are currently without evidence of disease
  * have not received treatment for invasive malignancy in the last 6 months
  * have no current or planned therapy, and
  * have an expected disease-free survival of at least 5 years from study entry
* Chronic use of: itraconazole; ketoconazole; erythromycin; clarithromycin; telithromycin; human immunodeficiency virus (HIV) protease inhibitors; nefazodone; cyclosporine; gemfibrozil and other fibrates; danazol; amiodarone (amiodarone hydrochloride); verapamil; coumarin anticoagulants; niacin (nicotinic acid) (>= 1 g/day); or large quantities of grapefruit juice (> l quart daily)
* Subjects with a history of coronary artery disease or stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-05; Primary Completion 2011-04 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Linden, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (3):
- United States (3):
  - University of California Medical Center At Irvine-Orange Campus, Orange, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Huntsman Cancer Institute, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Two Matched Nevi Group - Lovastatin | Two Matched Nevi Group - Placebo | One Large Nevi Group - Lovastatin | One Large Nevi Group - Placebo
Started | 34 | 32 | 7 | 7
Completed | 24 | 25 | 7 | 4
Not Completed | 10 | 7 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Two Matched Nevi Group-Lovastatin: Patients with two matched nevi received lovastatin PO QD for up to 6 months in the absence of disease progression or unacceptable toxicity.
  lovastatin: Given PO
  biopsy: Correlative studies
  laboratory biomarker analysis: Correlative studies
- Two Matched Nevi Group-Placebo: Patients with two matched nevi received placebo PO QD for up to 6 months in the absence of disease progression or unacceptable toxicity.
  placebo: Given PO
  biopsy: Correlative studies
  laboratory biomarker analysis: Correlative studies
- One Large Nevi Group-Lovastatin: Patients with one large nevi received placebo PO QD for up to 6 months in the absence of disease progression or unacceptable toxicity.
  lovastatin: Given PO
  biopsy: Correlative studies
  laboratory biomarker analysis: Correlative studies
- One Large Nevi Group-Placebo: Patients with one large nevi received placebo PO QD for up to 6 months in the absence of disease progression or unacceptable toxicity.
  placebo: Given PO
  biopsy: Correlative studies
  laboratory biomarker analysis: Correlative studies
- Total: Total of all reporting groups
Arm/Group | Two Matched Nevi Group-Lovastatin | Two Matched Nevi Group-Placebo | One Large Nevi Group-Lovastatin | One Large Nevi Group-Placebo | Total
Number analyzed (Participants) | 34 | 32 | 7 | 7 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.82 (10.96) | 42.16 (11.28) | 45.71 (10.98) | 36.29 (11.98) | 42.24 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 2 | 2 | 45
  Male | 13 | 12 | 5 | 5 | 35
Region of Enrollment [Number; unit: participants]
  United States | 34 | 32 | 7 | 7 | 80

OUTCOME MEASURES:

1. Primary Outcome: Histopathologic Regression of Target Atypical Nevi With Treatment - Pathologist 1's Evaluation
Description: The level of atypia will be graded in a standard fashion which leads to seven levels of atypia, with zero being no atypia and six being a melanoma. For each patient, the change from baseline in the level of atypia was calculated. Only the Two Matched Nevi Group - Lovastatin and Two Matched Nevi Group - Placebo data were used and analyzed for the primary outcome. One-Large Nevi Group - Lovastatin and One-Large Nevi Group - Placebo sample data were not used or analyzed due to insufficient numbers.
Time Frame: From baseline up to 24 weeks
Population: Only the Two Matched Nevi Group - Lovastatin and Two Matched Nevi Group - Placebo data were used and analyzed for the primary outcome. One-Large Nevi Group - Lovastatin and One-Large Nevi Group - Placebo sample data were not used or analyzed due to insufficient numbers.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Two Matched Nevi Group - Lovastatin | Two Matched Nevi Group - Placebo
Number analyzed (Participants) | 24 | 25
score | 0.50 (1.10) | -0.12 (1.33)

2. Secondary Outcome: Clinical Regression of Atypical Moles - Average of Three Reviewers' Evaluations
Description: From close-up photos of target atypical nevi, lesions will be graded clinically. After unblinding of pre- or post-treatment status for photos, the grading score was as follows: 1= Post-treatment (Post-TX) photo shows a complete resolution of atypia relative to pre-treatment (Pre-TX) photo, 2 = Post-TX photo shows a strong lessening of atypia relative to Pre-TX photo, 3 = Post-TX photo shows a mild lessening of atypia relative to Pre-TX photo, 4 = Post-TX and Pre-TX photos show same degree of atypia, 5 = Pre-TX photo shows a mild lessening of atypia relative to Post-TX photo, 6 = Pre-TX photo shows a strong lessening of atypia relative to Post-TX photo, 7 = Pre-TX photo shows a complete resolution of atypia relative to Post-TX photo. The Wilcoxon rank sum test will be applied to compare the scores for patients treated with placebo vs. those treated with lovastatin.
Time Frame: From baseline up to 24 weeks
Population: One Large Nevi Group-Lovastatin and Two Matched Nevi Group-Lovastatin arms are combined into the "Lovastatin" arm while One Large Nevi Group-Placebo and Two Matched Nevi Group-Placebo arms are combined into the "Placebo" arm. The total number of participants who have complete data are analyzed in this outcome measure.
Measure: Mean (Standard Deviation); unit: score
Groups:
- Lovastatin: One Large Nevi Group-Lovastatin and Two Matched Nevi Group-Lovastatin arms are combined into the "Lovastatin" arm. Patients received lovastatin PO QD for up to 6 months in the absence of disease progression or unacceptable toxicity.
  lovastatin: Given PO
  biopsy: Correlative studies
  laboratory biomarker analysis: Correlative studies
- Placebo: One Large Nevi Group-Placebo and Two Matched Nevi Group-Placebo arms are combined into the "Placebo" arm. Patients received placebo PO QD for up to 6 months in the absence of disease progression or unacceptable toxicity
  placebo: Given PO
  biopsy: Correlative studies
  laboratory biomarker analysis: Correlative studies
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 20 | 27
score | 4.03 (0.26) | 3.98 (0.31)
Statistical Analysis 1: Comparison: Lovastatin vs Placebo; Test type: Superiority or Other; p = 0.61, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Total Nevus Number on Patient's Back - Combined Three Reviewers' Evaluations
Description: Assessed by photos of subjects' back pre and post treatment. These photos will be used to count, by blinded evaluators, the number of nevi on the back pre and post therapy.
Time Frame: From baseline up to 24 weeks
Population: as for outcome 2
Measure: Number; unit: pairs of photos
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 23 | 26
pairs of photos
  Fewer nevi after the treatment | 4 | 3
  Same number of nevi after treatment | 64 | 67
  More nevi after the treatment | 1 | 7

4. Secondary Outcome: Serum and Molecular Biomarkers - HIF1alpha: Pathologist 3's Evaluation
Description: HIF1alpha expression was assessed via nuclear staining, and the change in the percentage of positive stained cells from baseline to 24 weeks is calculated.
Time Frame: From baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percentage of cells that are positive
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 21 | 25
percentage of cells that are positive | 0.05 [-0.13 to 0.22] | -0.32 [-0.75 to 0.11]

5. Secondary Outcome: Serum and Molecular Biomarkers - (e)-Cadherin: Pathologist 3's Evaluation
Description: (e)-cadherin expression was assessed via cytoplasmic staining, and the change in the percentage of positive stained cells from baseline to 24 weeks is calculated.
Time Frame: From baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percentage of cells that are positive
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 15 | 19
percentage of cells that are positive | 0.67 [-7.29 to 8.63] | -7.37 [-20.60 to 5.86]

6. Primary Outcome: Histopathologic Regression of Target Atypical Nevi With Treatment - Pathologist 2's Evaluation
Description: as for outcome 1
Time Frame: From baseline up to 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Two Matched Nevi Group - Lovastatin | Two Matched Nevi Group - Placebo
Number analyzed (Participants) | 24 | 25
score | 0.17 (1.81) | 0.04 (1.95)

7. Secondary Outcome: Serum and Molecular Biomarkers - (n)-Cadherin: Pathologist 3's Evaluation
Description: (n)-cadherin expression was assessed via cytoplasmic staining, and the change in the percentage of positive stained cells from baseline to 24 weeks is calculated.
Time Frame: From baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percentage of cells that are positive
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 11 | 18
percentage of cells that are positive | 5.91 [-15.85 to 27.67] | -9.17 [-20.74 to 2.41]

8. Secondary Outcome: Serum and Molecular Biomarkers - VEGF: Pathologist 3's Evaluation
Description: VEGF expression was assessed via cytoplasmic staining, and the change in the percentage of positive stained cells from baseline to 24 weeks is calculated.
Time Frame: From baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percentage of cells that are positive
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 16 | 19
percentage of cells that are positive | 4.81 [-11.92 to 21.55] | -0.63 [-17.89 to 16.63]

9. Secondary Outcome: Serum and Molecular Biomarkers - RelA: Pathologist 3's Evaluation
Description: RelA expression was assessed via cytoplasmic staining, and the change in the percentage of positive stained cells from baseline to 24 weeks is calculated.
Time Frame: From baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percentage of cells that are positive
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 12 | 16
percentage of cells that are positive | 0.83 [-1.00 to 2.67] | -1.25 [-6.26 to 3.76]

10. Secondary Outcome: Serum and Molecular Biomarkers - p21 (WAF1/CIP1): Pathologist 3's Evaluation
Description: p21 expression was assessed via nuclear staining, and the change in the percentage of positive stained cells from baseline to 24 weeks is calculated.
Time Frame: From baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percentage of cells that are positive
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 10 | 17
percentage of cells that are positive | 1.00 [-13.09 to 15.09] | 1.18 [-10.59 to 12.94]

11. Secondary Outcome: Serum and Molecular Biomarkers - Ki-67: Pathologist 3's Evaluation
Description: Ki-67 expression was assessed via nuclear staining, and the change in the percentage of positive stained cells from baseline to 24 weeks is calculated.
Time Frame: From baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percentage of cells that are positive
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 15 | 20
percentage of cells that are positive | 0.73 [-1.48 to 2.94] | 0.50 [-0.39 to 1.39]

12. Secondary Outcome: Serum and Molecular Biomarkers - HIF1alpha: Pathologist 4's Evaluation
Description: as for outcome 4
Time Frame: From baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percentage of cells that are positive
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 23 | 25
percentage of cells that are positive | -0.04 [-0.13 to 0.05] | -0.04 [-0.12 to 0.04]

13. Secondary Outcome: Serum and Molecular Biomarkers - (e)-Cadherin: Pathologist 4's Evaluation
Description: as for outcome 5
Time Frame: From baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percentage of cells that are positive
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 22 | 25
percentage of cells that are positive | 4.23 [-6.72 to 15.17] | -7.40 [-20.10 to 5.30]

14. Secondary Outcome: Serum and Molecular Biomarkers - (n)-Cadherin: Pathologist 4's Evaluation
Description: as for outcome 7
Time Frame: From baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percentage of cells that are positive
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 21 | 25
percentage of cells that are positive | 4.24 [-11.64 to 20.11] | -3.52 [-9.45 to 2.41]

15. Secondary Outcome: Serum and Molecular Biomarkers - VEGF: Pathologist 4's Evaluation
Description: as for outcome 8
Time Frame: From baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percentage of cells that are positive
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 23 | 25
percentage of cells that are positive | -1.83 [-8.08 to 4.43] | -2.24 [-10.10 to 5.62]

16. Secondary Outcome: Serum and Molecular Biomarkers - RelA: Pathologist 4's Evaluation
Description: as for outcome 9
Time Frame: From baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percentage of cells that are positive
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 22 | 25
percentage of cells that are positive | 3.73 [-2.34 to 9.79] | -3.44 [-10.98 to 4.10]

17. Secondary Outcome: Serum and Molecular Biomarkers - p21 (WAF1/CIP1): Pathologist 4's Evaluation
Description: as for outcome 10
Time Frame: From baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percentage of cells that are positive
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 20 | 23
percentage of cells that are positive | 2.05 [-3.48 to 7.58] | -0.13 [-3.42 to 3.16]

18. Secondary Outcome: Serum and Molecular Biomarkers - Ki-67: Pathologist 4's Evaluation
Description: as for outcome 11
Time Frame: From baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: percentage of cells that are positive
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 21 | 25
percentage of cells that are positive | 0.57 [-0.81 to 1.96] | 0.28 [-0.43 to 0.99]

19. Secondary Outcome: Change in Cholesterol (mg/dL) From Baseline After Treatment
Time Frame: Baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/dL
Groups:
- Placebo: One Large Nevi Group-Placebo and Two Matched Nevi Group-Placebo arms are combined into the "Placebo" arm. Patients received placebo PO QD for up to 6 months in the absence of disease progression or unacceptable toxicity.
  placebo: Given PO
  biopsy: Correlative studies
  laboratory biomarker analysis: Correlative studies
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 28 | 26
mg/dL | -27.25 [-38.32 to -16.18] | -3.77 [-16.43 to 8.9]

20. Secondary Outcome: Change in LDL (mg/dL) From Baseline After Treatment
Time Frame: Baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 25 | 27
mg/dL | -25.28 [-35.6 to -14.96] | -0.4 [-12.54 to 11.74]

21. Secondary Outcome: Change in HDL (mg/dL) From Baseline After Treatment
Time Frame: Baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 24 | 27
mg/dL | -1.42 [-5.19 to 2.36] | -2.63 [-8.34 to 3.08]

22. Secondary Outcome: Change in Triglycerides (mg/dL) From Baseline After Treatment
Time Frame: Baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 28 | 26
mg/dL | 1.21 [-8.67 to 11.1] | 1.65 [-20.3 to 23.61]

23. Secondary Outcome: Change in SGOT/AST (U/L) From Baseline After Treatment
Time Frame: Baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 31 | 28
U/L | 3.42 [-0.73 to 7.57] | -0.75 [-3.43 to 1.93]

24. Secondary Outcome: Change in SGOT/ALT (U/L) From Baseline After Treatment
Time Frame: Baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 28 | 27
U/L | 5.61 [-0.5 to 11.72] | 2.93 [-1.17 to 7.02]

25. Secondary Outcome: Change in CPK (U/L) From Baseline After Treatment
Time Frame: Baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 31 | 29
U/L | 20.94 [-2.21 to 44.08] | 9.1 [-18.76 to 36.96]

26. Secondary Outcome: Change in C-reactive Protein (mg/dL) From Baseline After Treatment
Time Frame: Baseline up to 24 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 25 | 23
mg/dL | -0.3 [-0.96 to 0.37] | -0.11 [-0.26 to 0.03]

27. Secondary Outcome: At Least 1 Study-related Adverse Event Reported During the Study
Description: All participants will be evaluable for toxicity from the time of their informed consent. Incidence of adverse events graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0.
Time Frame: Baseline up to 26 weeks
Population: One Large Nevi Group-Lovastatin and Two Matched Nevi Group-Lovastatin arms are combined into the "Lovastatin" arm while One Large Nevi Group-Placebo and Two Matched Nevi Group-Placebo arms are combined into the "Placebo" arm.
Measure: Number; unit: participants
Arm/Group | Lovastatin | Placebo
Number analyzed (Participants) | 41 | 39
participants
  Yes | 14 | 11
  No | 27 | 28

ADVERSE EVENTS:
Time Frame: The onset date of adverse event is between the randomization date and the date of off-study.
Groups:
- Two Matched Nevi Group-Placebo: Patients receive placebo PO QD for up to 6 months in the absence of disease progression or unacceptable toxicity.
  placebo: Given PO
  biopsy: Correlative studies
  laboratory biomarker analysis: Correlative studies
- One Large Nevi Group-Lovastatin: Patients who have one large nevi received lovastatin PO QD for up to 6 months
- One Large Nevi Group-Placebo: Patients who have one large nevi receive placebo PO QD for up to 6 months
Arm/Group | Two Matched Nevi Group-Lovastatin | Two Matched Nevi Group-Placebo | One Large Nevi Group-Lovastatin | One Large Nevi Group-Placebo
Serious Adverse Events (participants affected / at risk) | 1/34 | 2/32 | 0/7 | 1/7
Other Adverse Events (participants affected / at risk) | 27/34 | 25/32 | 4/7 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Two Matched Nevi Group-Lovastatin (N=34) | Two Matched Nevi Group-Placebo (N=32) | One Large Nevi Group-Lovastatin (N=7) | One Large Nevi Group-Placebo (N=7)
ELEVATED CPK (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERBILIRUBINEMIA (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ROTATOR CUFF SURGERY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Two Matched Nevi Group-Lovastatin (N=34) | Two Matched Nevi Group-Placebo (N=32) | One Large Nevi Group-Lovastatin (N=7) | One Large Nevi Group-Placebo (N=7)
3 NEW MOLES (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACID REFLUX (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALT SGPT (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ARMS TINGLING AT NIGHT (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
AST SGOT (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ATYPICAL MOLE BIOPSY (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BIOPSY SITE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLADDER INFECTION (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
BLOATING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BREAST TENDERNESS (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COLD (General disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
COLD SORE OUTBREAK (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COLD SYMPTOMS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COLD-FEVER (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
COLPOSCOPY-STOMACH DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COMMON COLD (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 3 (4) | 1 (2) | 2 (3) | 0 (0)
CONSTIPATION( INTERMITTANT) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
CPK (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CRAMPS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DECREASED LIBIDO (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 4 (6) | 7 (10) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 5 (7) | 4 (6) | 0 (0) | 0 (0)
DIZZINESS - INTERMITTENT - 2-3 TIMES A WEEK (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DRY FINGER TIPS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ELEVATED BILIRUBIN LEVEL (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ELEVATED CPK (Investigations) | 3 (3) | 3 (4) | 0 (0) | 0 (0)
ELEVATED CREATINE KINASE (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ELEVATED LDH (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ELEVATED TOTAL CK (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ELEVATED TRIGLYCERIDES (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
EXTRA URINE (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FACELIFT (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 5 (7) | 6 (8) | 0 (0) | 1 (1)
FEVER (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FEVER SORE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FIBROIDS (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FLU (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
FLU-FEVER (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GAS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 8 (12) | 9 (15) | 1 (5) | 2 (2)
HEARTBURN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HIGH BLOOD PRESSURE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HIGH CHOLESTEROL LEVEL (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HIVES (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INDIGESTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 4 (6) | 4 (4) | 1 (1) | 0 (0)
INTERMITTENT INSOMNIA (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INTERMITTENT NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ITCHY AT BIOPSY SITE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ITCHY HAND (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
JOINT PAIN (Musculoskeletal and connective tissue disorders) | 3 (5) | 4 (5) | 0 (0) | 0 (0)
JOINT/BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
KIDNEY INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LEFT HIP PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LEFT HIP SENSITIVITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LIGHTHEADEDNESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LOOSE STOOLS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LOWER BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MENSTRUAL CRAMPS (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MOLE CHANGE, FATTER AND LIGHTER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MOLE ON NECK CHANGE IN APPEARANCE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MOLE REMOVAL (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
MOLES (2) BIOPSIED (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MOTION SICKNESS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MOUTH ULCERS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCLE ACHE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCLE CRAMPS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
MUSCLE CRAMPS/PAIN (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
MUSCLE PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 1 (1) | 0 (0)
MUSCLE PAIN - NECK, BACK, SHOULDER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCLE PAIN AND ACHES; (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCLE TWITCHES IN THE UPPER LEFT ARM (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 6 (7) | 10 (14) | 1 (1) | 0 (0)
NECK PAIN-ARTHRITIC (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEW FOOT PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NUMBNESS AND SHOOTING PAIN IN LOWER BACK AND LEGS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NUMBNESS AND TINGLING IN THE RIGHT ARM (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PAIN IN BREASTS (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PAIN LOWER BACK (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PAIN-SHOULDER MUSCLE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERIPHERAL NERVOUS SYSTEM ( PARESTHESIA) TINGLING SKIN- LEFT SIDE FACE. (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PHARYNIGITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNS LEFT HAND PARESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PULLED BACK - LUMBAR SPINE INJURY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULLED TENDON (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
RIB PAIN - INTERMITTENT (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RIGHT HIP PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RIGHT KNEE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RIGHT LEG WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ROOT CANAL (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SCALY MOLE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEBORRHEIC KERATOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SHINGLES (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SINUS INFECTION (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
SKIN CHANGES (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN REACTION TO BANDAID ADHESIVE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN TAG CHANGE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SLIGHTLY ATYPICAL LENTIGO (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SOFT STOOLS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SORE BACK (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SORE CALF MUSCLES (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
SPRAINED FINGER-PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
STOMACH ACHE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
STOMACH DISCOMFORT (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
STOMACH PAIN (Gastrointestinal disorders) | 4 (4) | 4 (5) | 1 (2) | 0 (0)
STOMACH UPSET (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
STOMACH UPSET/GASTROENTERITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
STREP THROAT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
SUNBURN (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
SWOLLEN ANKLE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TEETH SENSITIVITY (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
THYROID CANCER (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TINGLING IN R PALM (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TINGLING IN R THUMB & R INDEX (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TINGLING IN THE FEET (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TIRED (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TOOTH PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UNKNOWN CHANGE IN THE CERVICAL LYMPH NODE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UNKNOWN PERIPHERAL NERVOUS SYSTEM (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URI (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VISUAL DISTURBANCES (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
WISDOM TEETH EXTRACTION - TOOTH PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
YEAST INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less